CLINICAL TRIAL: NCT05187156
Title: Assessing and Enhancing Social Support to Improve Treatment Outcomes Among Veterans With PTSD (CDA 19-208)
Brief Title: Assessing and Enhancing Social Support
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI has transitioned to working outside of the VA - study will not continue
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDX 22-004; CDA 19-208 (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Stress Disorders, Post-Traumatic; Social Support
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Veterans will participate in a novel intervention to improve PTSD and social support
  Interventions: Behavioral: Behavioral Activation and Social Engagement
- Treatment as usual (Active Comparator): Veterans will participate in usual care in PCMHI
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Behavioral Activation and Social Engagement — brief, PCMHI-based psychotherapy using behavioral activation principles and focused attention on enhancement of social support
  Arms: Intervention
Behavioral: Treatment as usual — treatment as usual in PCMHI includes participation in any other skills-based groups or brief individual psychotherapy and medication management offered in PCMHI
  Arms: Treatment as usual

SUMMARY:
Posttraumatic stress disorder (PTSD) is a common and impairing problem among Veterans, many of whom first seek treatment in primary care settings. PTSD is linked to reduced quality of life and increased rates of suicide. Additionally, social support, defined as the availability of others to provide emotional or practical support when needed, is frequently poor for Veterans with PTSD. For Veterans with PTSD, poor social support negatively impacts PTSD treatment engagement and outcomes, interfering with PTSD recovery. There is a need for additional brief, primary care-based treatments for PTSD that also work to improve social support in traumatized Veterans. The proposed research seeks to evaluate and refine such an intervention and establish a protocol for routinely measuring social support to inform treatment. This intervention and measurement protocol will likely improve Veterans' mental health and social relationships.

DETAILED DESCRIPTION:
Background: PTSD is a significant problem for Veterans, most of whom are initially treated for posttraumatic stress disorder (PTSD) in Primary Care Mental Health Integration (PCMHI). Poor social support in this population is a risk factor for suicidal ideation, all-cause mortality, and worse treatment engagement and response. Preliminary research shows that approximately 60% of Veterans with PTSD present to specialty care intake appointments with poor social support. However, none of the existing PCMHI-based treatments for PTSD explicitly focus on social support generation or reengagement. Moreover, although the limited existing research suggests that the routine assessment of social support to guide treatment planning (also known as measurement-based care, or MBC) improves treatment outcomes in civilian populations, social support is not routinely monitored as part of evidence-based treatments for PTSD. Thus, this CDA-2 will first identify an appropriate instrument for routinely measuring social support in the context of clinical care to improve PTSD treatment, and, subsequently, evaluate a novel PCMHI-based PTSD treatment as part of a stepped care model for Veterans who report poor social support and are at great risk of PTSD treatment non-response. Significance/Impact: The proposed research addresses several HSR&D research priorities, including evaluating the impact of social determinants of health, namely, social support, on the quality and outcomes of care; testing new models of mental health care to improve outcomes; and intervening with vulnerable Veterans with PTSD and suicide risk. By measuring and improving social support to enhance PTSD treatment, the proposed research plan explicitly addresses a key factor that impedes treatment outcomes for a sensitive population of Veterans. Innovation: Although poor social support is widely recognized as among the strongest predictors of PTSD development and maintenance, none of the existing PCMHI-based treatments for PTSD target or measure social support as a primary treatment focus. The proposed CDA-2 research is thus highly novel. No past or present HSR&D-funded studies have tested methods for monitoring or improving social support in PCMHI-based treatment among Veterans with PTSD, despite its association with poor clinical outcomes. Specific Aims: 1) Select an instrument for MBC of social support in clinical settings for Veterans with PTSD. 2) Iteratively refine and conduct a one-arm pilot test a brief, PCMHI-based behavioral activation and social engagement intervention for PTSD based on key stakeholder (e.g., Veteran and PCMHI provider) feedback. 3) Conduct a two-arm pilot randomized clinical trial (RCT) comparing the intervention to usual care in PCMHI. Methodology: Aim 1 will use quantitative data gathered in an online survey from 210 Veterans to assess the degree to which four measures of social support (identified via systematic review and clinical utility ranking) are acceptable, reliable, and sensitive, and select the best measure for use in Aim 2's pilot. Aim 2 will involve the iterative refinement of the PTSD and social support intervention following, and followed by, qualitative interviews with key stakeholders. Aim 2 will obtain data on participant acceptability, provider fidelity, and social-support-related MBC. The pilot RCT comparing the social support and PTSD intervention to usual care in Aim 3 will evaluate the feasibility and acceptability of recruitment, randomization, intervention engagement, evaluation strategy, and outcome measurement of clinical outcomes (e.g., PTSD, depression symptoms, and social support), as well as mechanisms of change (e.g., disclosure) and multiple stepped-care outcomes (e.g., clinically-indicated evidence-based psychotherapy initiation/retention). Next Steps/Implementation: This work will support future trials establishing effectiveness and implementation potential of the intervention, as well as a model of MBC of social support. Future research will explore MBC and PCMHI-based interventions for poor social support in related conditions.

ELIGIBILITY:
Inclusion Criteria:

Veterans will be eligible for participation if they:

* are currently enrolled in a Primary Care Clinic at VA Puget Sound Health Care System (VAPSHCS) (including Women's Clinic) or VAPSHCS Primary Care Mental Health Integration (PCMHI)
* meet criteria for clinical or subclinical PTSD consistent with PTSD treatment in PCMHI defined as > 33 on the PTSD Checklist for DSM 5 (PCL-5)
* are willing to have therapy sessions audiotaped for the purposes of fidelity assessment
* plan to live in Washington state for 6 months following entry into the study to prevent delivery of care across state lines

Exclusion Criteria:

* presence of severe mental illness (e.g., active psychosis and/or bipolar disorder)
* a psychiatric in-patient admission in the past 30 days
* medical record suicide flag
* a behavioral flag in the medical record
* individuals with impaired decision making capacity (as measured by evidence in the medical record of moderate-severe TBI, uncontrolled psychosis, dementia, communication flag, or inability to provide informed consent)
* individuals who are illiterate or have limited or no English proficiency
* medication change in the last month
* current or recent (last 6 months) participation in specialty mental health
* current participation in CPT or PE, to ensure that Veterans are representative of PCMHI

Inclusion/exclusion criteria will be assessed via chart review.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Percent completing treatment | Up to 16 weeks
  number completing treatment/number enrolled (ratio of the two variables)

SECONDARY OUTCOMES:
Percentage declined participation | up to 16 weeks
  number enrolled/number approached (ratio of the two variables)
PTSD Checklist for DSM-5 | change from baseline to up to 20 weeks
  Scores range from 0-80 with lower scores indicating lower levels of symptoms
PROMIS Depression Short Form 8 | change from baseline to up to 20 weeks
  Scores range from 8-40 with lower scores indicating lower levels of symptoms
Change in social support | change from baseline to up to 20 weeks
  Instrument to be selected based on results of qualitative interviews
Interpersonal Needs Questionnaire - Thwarted Belongingness Subscale | change from baseline to up to 20 weeks
  Scores range from 10-70 with lower scores indicating higher levels of social connection

OTHER OUTCOMES:
Counts of outpatient mental health visits by type | number occurring between up to 16 weeks and up to 40 weeks
  Number of specialty care encounters including medication management and psychotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Sarah B Campbell, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No